CLINICAL TRIAL: NCT06802107
Title: The Effects of Forward and Backward Treadmill Walking Exercises in Addition to Conventional Physiotherapy on Pain, Physical Performance and Balance in Knee Osteoarthritis
Brief Title: Effects of Different Walking Exercises on Pain, Physical Performance and Balance in Knee Osteoarthritis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, TAHIR DEDEOGLU, phd student, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HasanKUTDEDEOGLU001
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; Walking; Treadmill; Backward; Forward
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Backward-treadmill Walking Group (Experimental): Individuals in this group will do backward treadmill walking in addition to traditional physiotherapy.
  Interventions: Behavioral: Backward-treadmill Walking; Other: Traditional physiotherapy
- Forward-treadmill Walking Group (Experimental): Individuals in this group will do forward treadmill walking in addition to traditional physiotherapy.
  .
  Interventions: Behavioral: Forward-treadmill Walking; Other: Traditional physiotherapy
- Control Group (Active Comparator): This group will receive standard traditional physiotherapy. Traditional physiotherapy is a treatment method that includes exercise training, hotpack, ultrasound and TENS (electrotherapy) applications.
  Interventions: Other: Traditional physiotherapy

INTERVENTIONS:
Behavioral: Backward-treadmill Walking — A backward walking program will be applied on the treadmill. To be done 3 times a week / 8 weeks. Before the walking exercises, 5 minutes of warm-up and 5 minutes of cool-down exercises will be performed. While walking on the treadmill, the participant can hold onto the railings. Each participant will start at the speed they choose and gradually increase their perceived exertion rate to 11-13 on the Borg scale, and it is planned to walk for 10 minutes in the first week and gradually for 20-30 minutes in the following weeks.
  Arms: Backward-treadmill Walking Group
Behavioral: Forward-treadmill Walking — A forward walking program will be applied on the treadmill. To be done 3 times a week / 8 weeks. Before the walking exercises, 5 minutes of warm-up and 5 minutes of cool-down exercises will be performed. While walking on the treadmill, the participant can hold onto the railings. Each participant will start at the speed they choose and gradually increase their perceived exertion rate to 11-13 on the Borg scale, and it is planned to walk for 10 minutes in the first week and gradually for 20-30 minutes in the following weeks.
  Arms: Forward-treadmill Walking Group
Other: Traditional physiotherapy — Traditional physiotherapy is a treatment method that includes exercise training, hotpack, ultrasound and TENS (electrotherapy) applications.
  To be done 3 times a week / 8 weeks. 20 min hotpack + 7 min ultrasound + 20 min TENS and knee osteoarthritis exercises (hip knee flexion extension, knee extension while sitting on a chair, quadriceps isometric exercise in the supine position, straight leg raise exercises) are planned to be applied in the clinic with the physiotherapist. The exercises are planned to be started with 5 repetitions in the first week and the intensity of the exercise is planned to be increased with 10 repetitions, 15 repetitions and 20 repetitions depending on the patient's tolerance.

SUMMARY:
The aim of this study is to investigate and compare the effects of forward and backward walking exercises on treadmill in addition to traditional physiotherapy interventions on pain, physical performance and balance in patients with knee osteoarthritis. Secondarily, it is aimed to investigate the effects of walking on spatio-temporal parameters, knee joint position sense, range of motion, quadriceps, hamstring and hip adductors muscle strength, Q angle, quality of life and kinesiophobia.

DETAILED DESCRIPTION:
Knee osteoarthritis is a common degenerative joint disease in the world and causes varying degrees of loss of function in individuals in terms of pain, physical performance and balance ability due to the wear and tear in the joint cartilage. Exercise practices play a critical role in the management of knee osteoarthritis and various types of exercises are used to alleviate the symptoms of the disease. One of the exercises used in this context is walking. Today, various modified or designed walking training programs such as walking on land/water, weight-supported walking, positive pressure walking, walking on a treadmill, walking forward-backward, and walking uphill can be applied in the rehabilitation of individuals with osteoarthritis.

Exercises done on a treadmill offer individuals the opportunity to exercise safely in a controlled environment. In addition, forward and backward walking exercises done on a treadmill have the potential to improve balance and coordination by activating different muscle groups. Such dynamic exercises can facilitate the daily activities of osteoarthritis patients and increase their physical activity levels.

Some biomechanical research results on backward walking in recent years are quite interesting. It is stated that the quadriceps muscle works more concentrically and isometrically while the eccentric load decreases during backward walking and can be used to increase and strengthen the stability of the knee. In addition, according to studies conducted in recent years, walking backwards is a useful strategy to reduce knee load compared to forward walking. In light of these findings, it is a walking exercise type that is thought to be more effective for knee osteoarthritis rehabilitation. However, although there are many studies on the effects of walking exercise in knee osteoarthritis rehabilitation, there are very few studies on backward walking in knee osteoarthritis. At the same time, it is unclear whether walking backwards provides an additional clinical benefit compared to walking forward in patients with knee osteoarthritis. In addition, there is no study comparing the effects of walking backwards and walking forward on the treadmill on pain, physical performance and balance, and there is a serious gap in the literature on this subject.

In light of this information in the literature, the primary purpose of this study is to investigate and compare the effects of walking forwards and backwards on the treadmill in patients with knee osteoarthritis on pain, physical performance and balance. Secondarily, the effects of gait on spatio-temporal parameters, knee joint position sense, range of motion, quadriceps, hamstring and hip adductors muscle strength, Q angle, quality of life and kinesiophobia will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with knee OA
* According to the Kellgren Lawrence scale, grade I-II-III knee OA
* VAS score above 3

Exclusion Criteria:

* Knee pain caused by other diseases (rheumatoid arthritis, gouty arthritis, etc.)
* History of lower extremity surgery
* Receiving physical therapy within the last 6 months
* A medical condition that prevents safe exercise
* Intra-articular injection (hyaluronic acid/steroid) application within the last 6 months
* Diabetic neuropathy
* Active and regular exercise,
* Not volunteering to participate in the study
* Patients with osteoporosis

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain | 8 weeks
  It will be evaluated with the visual analog scale (VAS). VAS consists of a horizontal 10 cm long line, where "0" (zero) indicates no pain and "10" indicates unbearable pain. The patient is asked to indicate where their condition fits on this line by drawing a line, putting a dot or pointing.
Physical Function and Performance Measures | 8 weeks
  Western Ontario and McMaster Üniversiteleri Osteoartrit İndeksi (WOMAC) WOMAC is a self-reported health status measure developed to assess pain, joint stiffness, and function in patients with hip and knee osteoarthritis. It questions patients on three separate clinical dimensions: pain, joint stiffness, and function. It contains a total of 24 questions. The three subdimensions that make up the scale can be scored individually or as a total. Higher scores represent worse pain, physical function, and stiffness.
Physical Function and Performance Measures | 8 weeks
  30 second Chair test A test that evaluates the patient's sit-to-stay activity, lower extremity strength and dynamic balance. The number of times the patient sits down and stands up in 30 seconds gives the test score.
Physical Function and Performance Measures | 8 weeks
  40 meter fast paced walk test This test evaluates the speed and direction change activity of short-distance walking, especially in individuals with hip and knee osteoarthritis.
Physical Function and Performance Measures | 8 weeks
  Stair climb test A test that evaluates the patient's stair climbing and descending activity, lower extremity strength and dynamic balance. Ideally, the desired time to go up and down 9 steps gives the result of the test.
Physical Function and Performance Measures | 8 weeks
  6 minute walk test A test that evaluates functional capacity in individuals. The test is performed in a closed and uncrowded space. The distance between the starting and finishing points in a closed space should be 30 meters on a flat surface. The distance an individual can walk in this area in 6 minutes is evaluated in meters. Before the test begins, the patient is rested and information about the test is given to the patient. The patient is asked to walk between the starting and finishing points at their own walking pace. The test is monitored with a stopwatch. The purpose of the test is to measure the maximum distance they can walk during this time
balance | 8 weeks
  Timed up and go test This test measures the dynamic balance and functional mobility. It is a test that measures the time in seconds for the individual to stand up from a standard chair (seat height of approximately 44 cm, arm height 65 cm), walk a distance of 3 meters, turn around and sit on the chair.
balance | 8 weeks
  Functional Reach Test A test developed to examine forward stability. During the test, participants' ability to reach forward while standing with their feet fixed is recorded as a distance and their balance performance is evaluated.

SECONDARY OUTCOMES:
knee joint position sense | 8 weeks
  Joint position sense (JPS) is evaluated by the angular difference between a repeatedly determined target position and the predicted position, and this is called absolute angular error. This method is a reliable technique for the knee joint. JPS is tested by actively finding the joint position that was previously taught passively. In the study, 60° knee flexion were determined as target angles. It is planned to use a universal goniometer for the test.
Knee Range of Motion Assessment | 8 weeks
  Knee flexion and extension will be measured with a universal goniometer.
Quadriceps, Hamstring and hip adduction strength | 8 weeks
  Isometric muscle strength will be assessed with a hand-held dynamometer.
Q açısı | 8 weeks
  It is planned to be measured with a universal goniometer. The pivot point of the goniometer is placed at the center of the patella, the fixed arm pointing to the tibia tuberosity and the movable arm pointing to the SIAS, and the angle between the line drawn from the SIAS to the middle of the patella and the two lines drawn from the middle of the patella to the tibia tuberosity is recorded.
Kinesiophobia | 8 weeks
  Tampa Kinesiophobia Scale It was developed to evaluate the kinesiophobia of individuals. The scale consists of 17 questions. When calculating the scale score, the scores of some questions are reversed and calculated. A high total score indicates that the individual has high kinesiophobia.
Quality of life | 8 weeks
  EUROQL 5d 5l The scale consists of two parts: the EQ-5D descriptive system and the EQ-VAS (visual analog scale).
Spatio-temporal variables of gait | 8 weeks
  Gaı̇t Analyzer application A smartphone-based application called "Gait Analyzer" will be used. It collects kinematic data of gait using smartphone technology and phone sensors. With this application, kinematic data of walking such as walking speed, cadence, step duration, step length, step length symmetry and step duration symmetry can be obtained. The smartphone is fixed to the region corresponding to the L3 proccesus spinosus of the patient with a suitable waist belt with velcro bandage. The patients are then asked to walk a distance of 20 meters at their natural gait and speed without walking aids and measurements are performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Şahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No